CLINICAL TRIAL: NCT02485912
Title: A Phase Ib Safety and Immunogenicity Clinical Trial of Heterologous Prime-boost Immunisation With ChAd3-EBO Z and MVA-EBO Z in Healthy Senegalese Adult Volunteers Aged 18-50 Years.
Brief Title: Evaluation of a New Ebola Vaccine Using a Short-interval Prime-boost Vaccination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Centre Hospitalier Universitaire le Dantec (CHUD), Dakar, Senegal (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EBL06
Record Dates: First submitted 2015-06-25; First posted 2015-06-30 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2016-02

CONDITIONS: Ebola Virus Disease
Keywords: Ebola; vaccine; safety; immunogenicity
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): ChAd3-EBO Z (2.5 - 3.7 x 10^10 vp) and MVA-EBO Z (1.0 x 10^8 pfu) 7 days later. Both vaccinations are administered in the same arm.
  Interventions: Biological: ChAd3-EBO Z; Biological: MVA-EBO Z
- Group 2 (Active Comparator): ChAd3-EBO Z (2.5 - 3.7 x 10^10 vp) and MVA-EBO Z (1.0 x 10^8 pfu) 7 days later. The MVA-EBO Z is administered in the opposite arm to the ChAd3-EBO Z.
  Interventions: Biological: ChAd3-EBO Z; Biological: MVA-EBO Z

INTERVENTIONS:
Biological: ChAd3-EBO Z — This is a viral vectored vaccine using a chimpanzee adenovirus as a vector encoding a Zaire strain Ebola glycoprotein
Biological: MVA-EBO Z — This is a viral vectored vaccine using a modified vaccinia Ankara virus as a vector encoding a Zaire strain Ebola virus glycoprotein

SUMMARY:
This is a clinical trial in which healthy volunteers will be administered two experimental Ebola vaccines: ChAd3-EBO Z and MVA-EBO Z. Two groups of volunteers will be vaccinated with both vaccines one after the other in a prime/boost regimen.

All ChAd3-EBO Z doses are 2.5 x 10^10 - 3.7 x 10^10 vp and all MVA-EBO Z doses are 1.0 x 10^8 pfu.

All volunteers will receive a ChAd3-EBO Z priming vaccine and a MVA-EBO Z boosting vaccine 7 days later.

The site of administration of the MVA-EBO Z vaccine differs between the two groups:

Group 1 will receive the MVA-EBO Z vaccine in the same arm as the ChAd3-EBO Z vaccine.

Group 2 will receive the MVA-EBO Z vaccine in the opposite arm from the ChAd3-EBO Z vaccine.

The study will assess the safety of the vaccinations, and the immune responses to vaccination. Immune responses are measured by tests on blood samples.

The ChAd3-EBO Z and MVA-EBO Z vaccines are called viral vectored vaccines. They are made from viruses which are modified so that they cannot multiply. The viruses have extra DNA in them so that after injection, the body makes Ebola proteins (but Ebola does not develop), so that the immune system builds a response to Ebola without having been infected by it.

Healthy volunteers will be recruited in Dakar, Senegal. The study will be funded by GSK.

DETAILED DESCRIPTION:
The CHUD study team will hold sensitisation meetings, in specific areas targeting specific populations, to explain the study to potential volunteers. During these meetings the investigators will explain the following: the need for a vaccine (including a simple picture of the burden of the Ebola disease and how it affects the community); the current status of vaccine development (including the fact that this is likely to be a prolonged process that probably will not influence the course of the current epidemic); the study screening and informed consent procedure; risks of vaccination and the unproven benefits of this vaccination. It will be stressed that this is an experimental vaccine and there is no current evidence that it will provide protection, and that it will therefore still be necessary to take preventive measures and to seek treatment if ill for any reason after vaccination.

After these sensitisation meetings, the CT team will actively identify. The study will be further explained to eligible participants on individual basis. Potential volunteers will be invited to the CHUD CT site for further discussion. Potential volunteers will be informed that they are free to withdraw from the CT at any time without giving any reason. Individuals who feel that the trial is appropriate for them will be invited to attend a formal screening visit.

Detailed information about the study will be provided in a Participant Information Sheet (PIS) at least 24 hours prior to the consent being undertaken. The informed consent process will start before the screening visit. The volunteer will be given the opportunity to ask about details of the trial, and will then have time to consider whether or not to participate. The investigators will ensure that the volunteers are briefed on the contents of the PIS in the language they understand. The investigators will also ensure that all volunteers fully understand the risks. Any volunteer who appears to have less than complete understanding will not be enrolled.

All volunteers will sign and date the informed consent form before any study specific procedures (including screening visit) are performed. If the volunteer is illiterate, s/he will sign the informed consent form; in the latter case a literate adult impartial witness will be present throughout the whole consenting process, write subject's name and date of signature and will sign and date the consent form. Volunteers will sign and date two copies of the consent form, one for them to take away and keep, and one to be stored in the subject's medical records.

Vaccinations in Group 1 can commence 7 days after vaccination after interim safety review of the first 5 volunteers receiving the same dose in the UK CT. The first 5 volunteers will be vaccinated in a staggered fashion.

The first volunteer to receive the ChAd63-EBO Z vaccine dose in Group 1 will be vaccinated alone and we will wait 24 hours before vaccinating subsequent volunteers in this group. Two further Group 1 volunteers will be vaccinated 24 hours after the first, and then at least another 24 hours gap will pass before vaccinating further subjects receiving the ChAd63-EBO Z vaccine in Groups 1 & 2.

The same staggered vaccine administration procedure will be adopted for vaccinations with the MVA-EBO Z vaccine. A total of 20 volunteers will be enrolled in this group.

In Group 2, vaccination can commence after 5 volunteers in Groups 1 have received the ChAd63-EBO Z vaccine dose. The same staggered vaccine administration procedure as for Group 1 will be adopted for vaccinations with the MVA-EBO Z vaccine. A total of 20 volunteers will be enrolled in this group.

Volunteers will be visited daily at home by a study field worker or nurse to record adverse events (solicited and unsolicited for six consecutive days after vaccination). Additional scheduled visits at the CHUD clinic will be at day 7, 14, 28, 35, 56, 90, 180 post-first vaccination during which interim history will be collected, physical examination and blood tests performed at the time-points indicated in the schedule of attendances. Blood will also be taken for exploratory immunology analysis.

All volunteers will be followed up for 6 months beginning from the day of the first vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* For females only, willingness to practice continuous effective contraception (see section 6.4.3) during the study and a negative pregnancy test on the day(s) of screening and vaccination
* Agreement to refrain from blood donation during the course of the study
* Provide written informed consent

Exclusion Criteria:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned participation during the study period
* Prior receipt of an investigational Ebola or Marburg vaccine, a chimpanzee adenovirus vectored vaccine, an MVA vaccine or any other investigational vaccine likely to impact on interpretation of the trial data
* Receipt of any live, attenuated vaccine within 28 days prior to enrolment
* Receipt of any subunit or killed vaccine within 14 days prior to enrolment
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, (e.g. egg products) including urticaria, respiratory difficulty or abdominal pain
* Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
* Any history of anaphylaxis in reaction to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of current or previous psychiatric illness.
* Poorly controlled asthma or thyroid disease
* Seizure in the past 3 years or treatment for seizure disorder in the past 3 years
* Bleeding disorder (eg. Factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
* Any other serious chronic illness
* Current anti-tuberculosis prophylaxis or therapy
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Seropositive for hepatitis B surface antigen (HBsAg)
* History of contact with suspected, probable or confirmed cases of Ebola in the previous 21 days
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis (see Appendix A & B)
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Souleymane Mboup, MD; PhD, Principal Investigator — Centre Hospitalier Universitaire le Dantec (CHUD), Dakar, Senegal
Locations (1):
- Centre Hospitalier Universitaire le Dantec, Dakar, Senegal

REFERENCES:
- [Background] Dixon MG, Schafer IJ; Centers for Disease Control and Prevention (CDC). Ebola viral disease outbreak--West Africa, 2014. MMWR Morb Mortal Wkly Rep. 2014 Jun 27;63(25):548-51. PMID 24964881
- [Background] Kuhn JH, Bao Y, Bavari S, Becker S, Bradfute S, Brister JR, Bukreyev AA, Chandran K, Davey RA, Dolnik O, Dye JM, Enterlein S, Hensley LE, Honko AN, Jahrling PB, Johnson KM, Kobinger G, Leroy EM, Lever MS, Muhlberger E, Netesov SV, Olinger GG, Palacios G, Patterson JL, Paweska JT, Pitt L, Radoshitzky SR, Saphire EO, Smither SJ, Swanepoel R, Towner JS, van der Groen G, Volchkov VE, Wahl-Jensen V, Warren TK, Weidmann M, Nichol ST. Virus nomenclature below the species level: a standardized nomenclature for natural variants of viruses assigned to the family Filoviridae. Arch Virol. 2013 Jan;158(1):301-11. doi: 10.1007/s00705-012-1454-0. Epub 2012 Sep 23. PMID 23001720
- [Background] Sanchez A, Kiley MP, Holloway BP, Auperin DD. Sequence analysis of the Ebola virus genome: organization, genetic elements, and comparison with the genome of Marburg virus. Virus Res. 1993 Sep;29(3):215-40. doi: 10.1016/0168-1702(93)90063-s. PMID 8237108
- [Background] Sanchez A, Kiley MP, Klenk HD, Feldmann H. Sequence analysis of the Marburg virus nucleoprotein gene: comparison to Ebola virus and other non-segmented negative-strand RNA viruses. J Gen Virol. 1992 Feb;73 ( Pt 2):347-57. doi: 10.1099/0022-1317-73-2-347. PMID 1538192
- [Background] Hart MK. Vaccine research efforts for filoviruses. Int J Parasitol. 2003 May;33(5-6):583-95. doi: 10.1016/s0020-7519(03)00064-x. PMID 12782057
- [Background] Geisbert TW, Jahrling PB. Exotic emerging viral diseases: progress and challenges. Nat Med. 2004 Dec;10(12 Suppl):S110-21. doi: 10.1038/nm1142. PMID 15577929
- [Background] Meslin FX. Global aspects of emerging and potential zoonoses: a WHO perspective. Emerg Infect Dis. 1997 Apr-Jun;3(2):223-8. doi: 10.3201/eid0302.970220. PMID 9204308
- [Background] Okware SI, Omaswa FG, Zaramba S, Opio A, Lutwama JJ, Kamugisha J, Rwaguma EB, Kagwa P, Lamunu M. An outbreak of Ebola in Uganda. Trop Med Int Health. 2002 Dec;7(12):1068-75. doi: 10.1046/j.1365-3156.2002.00944.x. PMID 12460399
- [Background] Hensley LE, Jones SM, Feldmann H, Jahrling PB, Geisbert TW. Ebola and Marburg viruses: pathogenesis and development of countermeasures. Curr Mol Med. 2005 Dec;5(8):761-72. doi: 10.2174/156652405774962344. PMID 16375711
- [Background] Sullivan N, Yang ZY, Nabel GJ. Ebola virus pathogenesis: implications for vaccines and therapies. J Virol. 2003 Sep;77(18):9733-7. doi: 10.1128/jvi.77.18.9733-9737.2003. No abstract available. PMID 12941881
- [Background] Martin JE, Sullivan NJ, Enama ME, Gordon IJ, Roederer M, Koup RA, Bailer RT, Chakrabarti BK, Bailey MA, Gomez PL, Andrews CA, Moodie Z, Gu L, Stein JA, Nabel GJ, Graham BS. A DNA vaccine for Ebola virus is safe and immunogenic in a phase I clinical trial. Clin Vaccine Immunol. 2006 Nov;13(11):1267-77. doi: 10.1128/CVI.00162-06. Epub 2006 Sep 20. PMID 16988008
- [Background] Ledgerwood JE, Costner P, Desai N, Holman L, Enama ME, Yamshchikov G, Mulangu S, Hu Z, Andrews CA, Sheets RA, Koup RA, Roederer M, Bailer R, Mascola JR, Pau MG, Sullivan NJ, Goudsmit J, Nabel GJ, Graham BS; VRC 205 Study Team. A replication defective recombinant Ad5 vaccine expressing Ebola virus GP is safe and immunogenic in healthy adults. Vaccine. 2010 Dec 16;29(2):304-13. doi: 10.1016/j.vaccine.2010.10.037. Epub 2010 Oct 27. PMID 21034824
- [Background] Yang ZY, Duckers HJ, Sullivan NJ, Sanchez A, Nabel EG, Nabel GJ. Identification of the Ebola virus glycoprotein as the main viral determinant of vascular cell cytotoxicity and injury. Nat Med. 2000 Aug;6(8):886-9. doi: 10.1038/78645. PMID 10932225
- [Background] Sullivan NJ, Geisbert TW, Geisbert JB, Shedlock DJ, Xu L, Lamoreaux L, Custers JH, Popernack PM, Yang ZY, Pau MG, Roederer M, Koup RA, Goudsmit J, Jahrling PB, Nabel GJ. Immune protection of nonhuman primates against Ebola virus with single low-dose adenovirus vectors encoding modified GPs. PLoS Med. 2006 Jun;3(6):e177. doi: 10.1371/journal.pmed.0030177. Epub 2006 May 16. PMID 16683867
- [Background] Bett AJ, Haddara W, Prevec L, Graham FL. An efficient and flexible system for construction of adenovirus vectors with insertions or deletions in early regions 1 and 3. Proc Natl Acad Sci U S A. 1994 Sep 13;91(19):8802-6. doi: 10.1073/pnas.91.19.8802. PMID 8090727
- [Background] Top FH Jr, Grossman RA, Bartelloni PJ, Segal HE, Dudding BA, Russell PK, Buescher EL. Immunization with live types 7 and 4 adenovirus vaccines. I. Safety, infectivity, antigenicity, and potency of adenovirus type 7 vaccine in humans. J Infect Dis. 1971 Aug;124(2):148-54. doi: 10.1093/infdis/124.2.148. No abstract available. PMID 4330997
- [Background] Tatsis N, Blejer A, Lasaro MO, Hensley SE, Cun A, Tesema L, Li Y, Gao GP, Xiang ZQ, Zhou D, Wilson JM, Ertl HC. A CD46-binding chimpanzee adenovirus vector as a vaccine carrier. Mol Ther. 2007 Mar;15(3):608-17. doi: 10.1038/sj.mt.6300078. Epub 2007 Jan 16. PMID 17228314
- [Background] Bruna-Romero O, Gonzalez-Aseguinolaza G, Hafalla JC, Tsuji M, Nussenzweig RS. Complete, long-lasting protection against malaria of mice primed and boosted with two distinct viral vectors expressing the same plasmodial antigen. Proc Natl Acad Sci U S A. 2001 Sep 25;98(20):11491-6. doi: 10.1073/pnas.191380898. Epub 2001 Sep 11. PMID 11553779
- [Background] Farina SF, Gao GP, Xiang ZQ, Rux JJ, Burnett RM, Alvira MR, Marsh J, Ertl HC, Wilson JM. Replication-defective vector based on a chimpanzee adenovirus. J Virol. 2001 Dec;75(23):11603-13. doi: 10.1128/JVI.75.23.11603-11613.2001. PMID 11689642
- [Background] Tatsis N, Tesema L, Robinson ER, Giles-Davis W, McCoy K, Gao GP, Wilson JM, Ertl HC. Chimpanzee-origin adenovirus vectors as vaccine carriers. Gene Ther. 2006 Mar;13(5):421-9. doi: 10.1038/sj.gt.3302675. PMID 16319951
- [Background] Barnes E, Folgori A, Capone S, Swadling L, Aston S, Kurioka A, Meyer J, Huddart R, Smith K, Townsend R, Brown A, Antrobus R, Ammendola V, Naddeo M, O'Hara G, Willberg C, Harrison A, Grazioli F, Esposito ML, Siani L, Traboni C, Oo Y, Adams D, Hill A, Colloca S, Nicosia A, Cortese R, Klenerman P. Novel adenovirus-based vaccines induce broad and sustained T cell responses to HCV in man. Sci Transl Med. 2012 Jan 4;4(115):115ra1. doi: 10.1126/scitranslmed.3003155. PMID 22218690
- [Background] O'Hara GA, Duncan CJ, Ewer KJ, Collins KA, Elias SC, Halstead FD, Goodman AL, Edwards NJ, Reyes-Sandoval A, Bird P, Rowland R, Sheehy SH, Poulton ID, Hutchings C, Todryk S, Andrews L, Folgori A, Berrie E, Moyle S, Nicosia A, Colloca S, Cortese R, Siani L, Lawrie AM, Gilbert SC, Hill AV. Clinical assessment of a recombinant simian adenovirus ChAd63: a potent new vaccine vector. J Infect Dis. 2012 Mar 1;205(5):772-81. doi: 10.1093/infdis/jir850. Epub 2012 Jan 24. PMID 22275401
- [Background] Colloca S, Barnes E, Folgori A, Ammendola V, Capone S, Cirillo A, Siani L, Naddeo M, Grazioli F, Esposito ML, Ambrosio M, Sparacino A, Bartiromo M, Meola A, Smith K, Kurioka A, O'Hara GA, Ewer KJ, Anagnostou N, Bliss C, Hill AV, Traboni C, Klenerman P, Cortese R, Nicosia A. Vaccine vectors derived from a large collection of simian adenoviruses induce potent cellular immunity across multiple species. Sci Transl Med. 2012 Jan 4;4(115):115ra2. doi: 10.1126/scitranslmed.3002925. PMID 22218691
- [Background] Peruzzi D, Dharmapuri S, Cirillo A, Bruni BE, Nicosia A, Cortese R, Colloca S, Ciliberto G, La Monica N, Aurisicchio L. A novel chimpanzee serotype-based adenoviral vector as delivery tool for cancer vaccines. Vaccine. 2009 Feb 25;27(9):1293-300. doi: 10.1016/j.vaccine.2008.12.051. Epub 2009 Jan 20. PMID 19162112
- [Background] Quinn KM, Da Costa A, Yamamoto A, Berry D, Lindsay RW, Darrah PA, Wang L, Cheng C, Kong WP, Gall JG, Nicosia A, Folgori A, Colloca S, Cortese R, Gostick E, Price DA, Gomez CE, Esteban M, Wyatt LS, Moss B, Morgan C, Roederer M, Bailer RT, Nabel GJ, Koup RA, Seder RA. Comparative analysis of the magnitude, quality, phenotype, and protective capacity of simian immunodeficiency virus gag-specific CD8+ T cells following human-, simian-, and chimpanzee-derived recombinant adenoviral vector immunization. J Immunol. 2013 Mar 15;190(6):2720-35. doi: 10.4049/jimmunol.1202861. Epub 2013 Feb 6. PMID 23390298
- [Background] Ledgerwood JE, DeZure AD, Stanley DA, Coates EE, Novik L, Enama ME, Berkowitz NM, Hu Z, Joshi G, Ploquin A, Sitar S, Gordon IJ, Plummer SA, Holman LA, Hendel CS, Yamshchikov G, Roman F, Nicosia A, Colloca S, Cortese R, Bailer RT, Schwartz RM, Roederer M, Mascola JR, Koup RA, Sullivan NJ, Graham BS; VRC 207 Study Team. Chimpanzee Adenovirus Vector Ebola Vaccine. N Engl J Med. 2017 Mar 9;376(10):928-938. doi: 10.1056/NEJMoa1410863. Epub 2014 Nov 26. PMID 25426834
- [Background] Ewer K, Rampling T, Venkatraman N, Bowyer G, Wright D, Lambe T, Imoukhuede EB, Payne R, Fehling SK, Strecker T, Biedenkopf N, Krahling V, Tully CM, Edwards NJ, Bentley EM, Samuel D, Labbe G, Jin J, Gibani M, Minhinnick A, Wilkie M, Poulton I, Lella N, Roberts R, Hartnell F, Bliss C, Sierra-Davidson K, Powlson J, Berrie E, Tedder R, Roman F, De Ryck I, Nicosia A, Sullivan NJ, Stanley DA, Mbaya OT, Ledgerwood JE, Schwartz RM, Siani L, Colloca S, Folgori A, Di Marco S, Cortese R, Wright E, Becker S, Graham BS, Koup RA, Levine MM, Volkmann A, Chaplin P, Pollard AJ, Draper SJ, Ballou WR, Lawrie A, Gilbert SC, Hill AV. A Monovalent Chimpanzee Adenovirus Ebola Vaccine Boosted with MVA. N Engl J Med. 2016 Apr 28;374(17):1635-46. doi: 10.1056/NEJMoa1411627. Epub 2015 Jan 28. PMID 25629663
- [Background] Mayr A, Stickl H, Muller HK, Danner K, Singer H. [The smallpox vaccination strain MVA: marker, genetic structure, experience gained with the parenteral vaccination and behavior in organisms with a debilitated defence mechanism (author's transl)]. Zentralbl Bakteriol B. 1978 Dec;167(5-6):375-90. German. PMID 219640
- [Background] Lohr V, Rath A, Genzel Y, Jordan I, Sandig V, Reichl U. New avian suspension cell lines provide production of influenza virus and MVA in serum-free media: studies on growth, metabolism and virus propagation. Vaccine. 2009 Aug 6;27(36):4975-82. doi: 10.1016/j.vaccine.2009.05.083. Epub 2009 Jun 14. PMID 19531390
- [Background] Jordan I, Vos A, Beilfuss S, Neubert A, Breul S, Sandig V. An avian cell line designed for production of highly attenuated viruses. Vaccine. 2009 Jan 29;27(5):748-56. doi: 10.1016/j.vaccine.2008.11.066. Epub 2008 Dec 9. PMID 19071186
- [Background] Goepfert PA, Elizaga ML, Sato A, Qin L, Cardinali M, Hay CM, Hural J, DeRosa SC, DeFawe OD, Tomaras GD, Montefiori DC, Xu Y, Lai L, Kalams SA, Baden LR, Frey SE, Blattner WA, Wyatt LS, Moss B, Robinson HL; National Institute of Allergy and Infectious Diseases HIV Vaccine Trials Network. Phase 1 safety and immunogenicity testing of DNA and recombinant modified vaccinia Ankara vaccines expressing HIV-1 virus-like particles. J Infect Dis. 2011 Mar 1;203(5):610-9. doi: 10.1093/infdis/jiq105. Epub 2011 Jan 31. PMID 21282192
- [Background] Howles S, Guimaraes-Walker A, Yang H, Hancock G, di Gleria K, Tarragona-Fiol T, Hayes P, Gilmour J, Bridgeman A, Hanke T, McMichael A, Dorrell L. Vaccination with a modified vaccinia virus Ankara (MVA)-vectored HIV-1 immunogen induces modest vector-specific T cell responses in human subjects. Vaccine. 2010 Oct 21;28(45):7306-12. doi: 10.1016/j.vaccine.2010.08.077. Epub 2010 Sep 16. PMID 20816902
- [Background] Scriba TJ, Tameris M, Mansoor N, Smit E, van der Merwe L, Isaacs F, Keyser A, Moyo S, Brittain N, Lawrie A, Gelderbloem S, Veldsman A, Hatherill M, Hawkridge A, Hill AV, Hussey GD, Mahomed H, McShane H, Hanekom WA. Modified vaccinia Ankara-expressing Ag85A, a novel tuberculosis vaccine, is safe in adolescents and children, and induces polyfunctional CD4+ T cells. Eur J Immunol. 2010 Jan;40(1):279-90. doi: 10.1002/eji.200939754. PMID 20017188
- [Background] Berthoud TK, Hamill M, Lillie PJ, Hwenda L, Collins KA, Ewer KJ, Milicic A, Poyntz HC, Lambe T, Fletcher HA, Hill AV, Gilbert SC. Potent CD8+ T-cell immunogenicity in humans of a novel heterosubtypic influenza A vaccine, MVA-NP+M1. Clin Infect Dis. 2011 Jan 1;52(1):1-7. doi: 10.1093/cid/ciq015. PMID 21148512
- [Background] Dangoor A, Lorigan P, Keilholz U, Schadendorf D, Harris A, Ottensmeier C, Smyth J, Hoffmann K, Anderson R, Cripps M, Schneider J, Hawkins R. Clinical and immunological responses in metastatic melanoma patients vaccinated with a high-dose poly-epitope vaccine. Cancer Immunol Immunother. 2010 Jun;59(6):863-73. doi: 10.1007/s00262-009-0811-7. Epub 2009 Dec 31. PMID 20043222
- [Background] Draper SJ, Heeney JL. Viruses as vaccine vectors for infectious diseases and cancer. Nat Rev Microbiol. 2010 Jan;8(1):62-73. doi: 10.1038/nrmicro2240. PMID 19966816
- [Background] Bejon P, Mwacharo J, Kai O, Mwangi T, Milligan P, Todryk S, Keating S, Lang T, Lowe B, Gikonyo C, Molyneux C, Fegan G, Gilbert SC, Peshu N, Marsh K, Hill AV. A phase 2b randomised trial of the candidate malaria vaccines FP9 ME-TRAP and MVA ME-TRAP among children in Kenya. PLoS Clin Trials. 2006 Oct 20;1(6):e29. doi: 10.1371/journal.pctr.0010029. PMID 17053830
- [Background] Moorthy VS, Imoukhuede EB, Milligan P, Bojang K, Keating S, Kaye P, Pinder M, Gilbert SC, Walraven G, Greenwood BM, Hill AS. A randomised, double-blind, controlled vaccine efficacy trial of DNA/MVA ME-TRAP against malaria infection in Gambian adults. PLoS Med. 2004 Nov;1(2):e33. doi: 10.1371/journal.pmed.0010033. Epub 2004 Oct 26. PMID 15526058
- [Background] Webster DP, Dunachie S, McConkey S, Poulton I, Moore AC, Walther M, Laidlaw SM, Peto T, Skinner MA, Gilbert SC, Hill AV. Safety of recombinant fowlpox strain FP9 and modified vaccinia virus Ankara vaccines against liver-stage P. falciparum malaria in non-immune volunteers. Vaccine. 2006 Apr 5;24(15):3026-34. doi: 10.1016/j.vaccine.2005.10.058. Epub 2006 Feb 2. PMID 16488059
- [Background] Sheehy SH, Duncan CJ, Elias SC, Biswas S, Collins KA, O'Hara GA, Halstead FD, Ewer KJ, Mahungu T, Spencer AJ, Miura K, Poulton ID, Dicks MD, Edwards NJ, Berrie E, Moyle S, Colloca S, Cortese R, Gantlett K, Long CA, Lawrie AM, Gilbert SC, Doherty T, Nicosia A, Hill AV, Draper SJ. Phase Ia clinical evaluation of the safety and immunogenicity of the Plasmodium falciparum blood-stage antigen AMA1 in ChAd63 and MVA vaccine vectors. PLoS One. 2012;7(2):e31208. doi: 10.1371/journal.pone.0031208. Epub 2012 Feb 21. PMID 22363582
- [Background] Sheehy SH, Duncan CJ, Elias SC, Collins KA, Ewer KJ, Spencer AJ, Williams AR, Halstead FD, Moretz SE, Miura K, Epp C, Dicks MD, Poulton ID, Lawrie AM, Berrie E, Moyle S, Long CA, Colloca S, Cortese R, Gilbert SC, Nicosia A, Hill AV, Draper SJ. Phase Ia clinical evaluation of the Plasmodium falciparum blood-stage antigen MSP1 in ChAd63 and MVA vaccine vectors. Mol Ther. 2011 Dec;19(12):2269-76. doi: 10.1038/mt.2011.176. Epub 2011 Aug 23. PMID 21862998
- [Background] Ogwang C, Afolabi M, Kimani D, Jagne YJ, Sheehy SH, Bliss CM, Duncan CJ, Collins KA, Garcia Knight MA, Kimani E, Anagnostou NA, Berrie E, Moyle S, Gilbert SC, Spencer AJ, Soipei P, Mueller J, Okebe J, Colloca S, Cortese R, Viebig NK, Roberts R, Gantlett K, Lawrie AM, Nicosia A, Imoukhuede EB, Bejon P, Urban BC, Flanagan KL, Ewer KJ, Chilengi R, Hill AV, Bojang K. Safety and immunogenicity of heterologous prime-boost immunisation with Plasmodium falciparum malaria candidate vaccines, ChAd63 ME-TRAP and MVA ME-TRAP, in healthy Gambian and Kenyan adults. PLoS One. 2013;8(3):e57726. doi: 10.1371/journal.pone.0057726. Epub 2013 Mar 19. PMID 23526949
- [Background] Sheehy SH, Duncan CJ, Elias SC, Choudhary P, Biswas S, Halstead FD, Collins KA, Edwards NJ, Douglas AD, Anagnostou NA, Ewer KJ, Havelock T, Mahungu T, Bliss CM, Miura K, Poulton ID, Lillie PJ, Antrobus RD, Berrie E, Moyle S, Gantlett K, Colloca S, Cortese R, Long CA, Sinden RE, Gilbert SC, Lawrie AM, Doherty T, Faust SN, Nicosia A, Hill AV, Draper SJ. ChAd63-MVA-vectored blood-stage malaria vaccines targeting MSP1 and AMA1: assessment of efficacy against mosquito bite challenge in humans. Mol Ther. 2012 Dec;20(12):2355-68. doi: 10.1038/mt.2012.223. Epub 2012 Oct 23. PMID 23089736
- [Background] Ewer KJ, O'Hara GA, Duncan CJ, Collins KA, Sheehy SH, Reyes-Sandoval A, Goodman AL, Edwards NJ, Elias SC, Halstead FD, Longley RJ, Rowland R, Poulton ID, Draper SJ, Blagborough AM, Berrie E, Moyle S, Williams N, Siani L, Folgori A, Colloca S, Sinden RE, Lawrie AM, Cortese R, Gilbert SC, Nicosia A, Hill AV. Protective CD8+ T-cell immunity to human malaria induced by chimpanzee adenovirus-MVA immunisation. Nat Commun. 2013;4:2836. doi: 10.1038/ncomms3836. PMID 24284865
- [Background] Sullivan NJ, Hensley L, Asiedu C, Geisbert TW, Stanley D, Johnson J, Honko A, Olinger G, Bailey M, Geisbert JB, Reimann KA, Bao S, Rao S, Roederer M, Jahrling PB, Koup RA, Nabel GJ. CD8+ cellular immunity mediates rAd5 vaccine protection against Ebola virus infection of nonhuman primates. Nat Med. 2011 Aug 21;17(9):1128-31. doi: 10.1038/nm.2447. PMID 21857654
- [Background] Malaeb BS, Gardner TA, Margulis V, Yang L, Gillenwater JY, Chung LW, Macik G, Koeneman KS. Elevated activated partial thromboplastin time during administration of first-generation adenoviral vectors for gene therapy for prostate cancer: identification of lupus anticoagulants. Urology. 2005 Oct;66(4):830-4. doi: 10.1016/j.urology.2005.04.041. PMID 16230147
- [Derived] Venkatraman N, Ndiaye BP, Bowyer G, Wade D, Sridhar S, Wright D, Powlson J, Ndiaye I, Dieye S, Thompson C, Bakhoum M, Morter R, Capone S, Del Sorbo M, Jamieson S, Rampling T, Datoo M, Roberts R, Poulton I, Griffiths O, Ballou WR, Roman F, Lewis DJM, Lawrie A, Imoukhuede E, Gilbert SC, Dieye TN, Ewer KJ, Mboup S, Hill AVS. Safety and Immunogenicity of a Heterologous Prime-Boost Ebola Virus Vaccine Regimen in Healthy Adults in the United Kingdom and Senegal. J Infect Dis. 2019 Apr 8;219(8):1187-1197. doi: 10.1093/infdis/jiy639. PMID 30407513

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 13 | 16 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Senegal | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Administration of ChAd3-EBO Z and MVA-EBO Z 7 Days Later. This Will be Done by Recording the Number of Participants Who Experience Adverse Events and the Severity of Any Adverse Events.
Description: The specific endpoints for safety and reactogenicity will be actively and passively collected data on adverse events.
  The following parameters will be assessed for both groups:
  * Occurrence of solicited local reactogenicity signs and symptoms for 7 days following the vaccination
  * Occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following the vaccination
  * Occurrence of unsolicited adverse events for 28 days following the vaccination
  * Change from baseline for safety laboratory measures
  * Occurrence of serious adverse events during the whole study duration
Time Frame: 26 weeks
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 20 | 20
participants | 20 | 20

2. Secondary Outcome: To Assess the Immunogenicity Generated by Heterologous Prime-boost Immunisation With Monovalent ChAd3-EBO Z (2.5 x 1010 vp - 3.7 x 1010vp) and MVA-EBO Z (1.0 x 108 Pfu) in Healthy Senegalese Volunteers Aged 18-50 Years
Description: Ebolavirus specific immunogenicity will be assessed by a variety of immunological assays. The primary immunogenicity outcome measures are ELISA and neutralization antigen-specific assays for antibody responses and intracellular cytokine staining (ICS) assay for T cell responses.
  Exploratory outcome measures will include ex-vivo ELISPOT, plasma blast assays and flow cytometry performed with research samples collected at different study timepoints as well as other immunogenicity assays throughout the study. An evaluation of genetic factors associated with immune responses may be performed as exploratory evaluation. Vaccine-induced mRNA expression profiles during 1 week after vaccination may also be performed as an exploratory evaluation.
Time Frame: 26 weeks
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 20 | 20
participants | 20 | 20

ADVERSE EVENTS:
Time Frame: Solicited adverse events will be recorded daily for 7 days post-vaccination Unsolicited AEs of all severities will be recorded from receipt of vaccination through 28 days post-vaccination. After study Day 28, only SAEs or new chronic medical conditions that require ongoing medical management will be recorded through to the last study visit.
Description: There was no serious adverse event.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 17/20 | 18/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=20) | Group 2 (N=20)
headache (Vascular disorders) | 8 (9) | 4 (4)
anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0)
Pain (General disorders) | 13 (18) | 10 (12)
warmth (General disorders) | 6 (6) | 1 (1)
itching (General disorders) | 4 (4) | 0 (0)
redness (General disorders) | 1 (1) | 1 (1)
myalgia (Nervous system disorders) | 5 (6) | 3 (3)
fatigue (General disorders) | 8 (9) | 2 (2)
nausea (General disorders) | 2 (3) | 0 (0)
malaise (General disorders) | 3 (3) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
neutropenia (Immune system disorders) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Feverish (General disorders) | 3 (3) | 0 (0)
Dysmenorrhea (General disorders) | 1 (1) | 0 (0)
feverish/chills (General disorders) | 1 (1) | 0 (0)
tooth pain (General disorders) | 1 (1) | 0 (0)
unwell (General disorders) | 1 (1) | 0 (0)
diarrhoea (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes